CLINICAL TRIAL: NCT00002827
Title: RESPONSE DEPENDENT TREATMENT OF STAGES IA, IIA AND IIIA HODGKIN'S DISEASE WITH DBVE AND LOW DOSE INVOLVED FIELD IRRADIATION WITH OR WITHOUT ZINECARD: A PEDIATRIC ONCOLOGY GROUP PHASE III STUDY
Brief Title: Chemotherapy Followed by Radiation Therapy in Treating Young Patients With Newly Diagnosed Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9426; POG-9426 (Other: Pediatric Oncology Group); CCG-P9426 (Other: Children's Cancer Group); CDR0000065013 (Other: Clinical Trials.gov); COG-9426 (Other: Children's Oncology Group)
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Cardiac Toxicity; Lymphoma
Keywords: stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; cardiac toxicity
MeSH Terms: conditions — Cardiotoxicity; Lymphoma | interventions — Bleomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; Vincristine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment #1 (Without Zinecard) (Experimental): All patients undergoing a splenectomy must receive penicillin or erythromycin prophylaxis twice a day. Pneumocystis prophylaxis:TMP/SMZ 150mg/m2(maximum 300 mg) of TMP in 2 divided doses on 3 consecutive days each week. Aerosolized Pentamidine (200mg/m2/dose - maximum dose 300 mg) should be substituted monthly for patients who cannot tolerate TMP/SMZ therapy. Continue pneumocystis prophylaxis for 6 months after stopping therapy.
  Doxorubicin hydrochloride 25mg/m2/day IV push over 15 minutes days 1 and 15 Bleomycin sulfate 10 IU/m2/day IV push over 10 minutes on days 1 and 15 Vincristine sulfate 1.5mg/m2/day IV push (maximum 2mg) days 1 and 15 Etoposide 10mg/m2/day 1-5. IV drip ( < 0.4mg/ml) over 1 hour. Monitor blood pressure every 15 minutes during infusion. G-CSF (filgrastim) 5 mcg/Kg/day start on day 6 (24-36 hrs after 5th dose of VP16) and continued through day 13 (total 8 days).
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy
- Treatment #2 (with Zinecard) (Experimental): Zinecard (DZR) 250 mg/m2 IV push on days 1 and 15 before administration of doxorubicin and bleomycin sulfate. Give bleomycin sulfate and doxorubicin within 30 minutes of Zinecard (dexrazoxane hydrochloride). Bleomycin 10 IU/m2/day IV push over 10 minutes on days 1 and 15 Doxorubicin hydrochloride 25mg/m2/day IV push over 15 minutes days 1 and 15 Vincristine Sulfate 1.5mg/m2/day IV push (maximum 2mg) days 1 and 15
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV
  Other Names: Blenoxane; NSC #125066
Biological: filgrastim — Given IV
  Other Names: Granulocyte-colony stimulating factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: dexrazoxane hydrochloride — Given IV
  Other Names: DZR; ADR-529; ZINECARD; ICRF-187; NSC #169780
  Arms: Treatment #2 (with Zinecard)
Drug: doxorubicin hydrochloride — Given IV
  Other Names: NSC #123127
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; NSC #141540
Drug: vincristine sulfate — Given IV
  Other Names: VCR; Oncovin; NSC #67574
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy with radiation therapy may kill more cancer cells. It is not yet known if chemotherapy is more effective with or without dexrazoxane for Hodgkin's disease.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy, with or without dexrazoxane, followed by radiation therapy in treating young patients with newly diagnosed stage I, stage II, or stage III Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Modify chemotherapy courses based on initial response to therapy in children with newly diagnosed stage IA/IIA/IIIA1 Hodgkin's disease. II. Examine the activity of variable courses of doxorubicin, bleomycin, vincristine, and etoposide (DBVE) followed by low-dose involved-field irradiation in these patients. III. Monitor the safety and feasibility of the response-dependent approach and the morbidity and immediate and long-term toxic effects associated with this regimen. IV. Assess whether limited therapy is adequate for patients with an early response. V. Evaluate whether the addition of dexrazoxane can reduce pulmonary toxicity while not significantly reducing the response rate or event-free survival. VI. Evaluate whether the frequency and magnitude of myocardial injury during therapy, as measured by elevated serum cardiac troponin-T, is reduced by the addition of dexrazoxane.

OUTLINE: This is a randomized study. Patients are stratified by participating institution. Patients are randomly assigned to receive doxorubicin, bleomycin, vincristine, etoposide, and filgrastim with vs. without dexrazoxane. Filgrastim SC begins on days 6-13; no filgrastim is given on day 14 or 15. Filgrastim will restart 2 days after completing therapy and continue until count recovery from expected nadir (ANC greater than 1000 cubic meter after nadir). Courses repeat every 28 days. Those with stable or responding disease after 2-4 courses receive involved-field radiotherapy 5 days per week for 3.5 weeks. Tanner stage IV/V patients are eligible for randomization based on a front-end institutional agreement and may receive standard-field radiotherapy 5 days per week for up to 11 weeks at the investigator's discretion. Patients are followed yearly until relapse, death, or for a minimum of 10 years.

PROJECTED ACCRUAL: A total of 285 patients will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Hodgkin's disease No more than 5 weeks since diagnostic biopsy No B symptoms Clinical/pathologic stages (all histologies) as follows: Stage IA/IIA with mediastinal mass less than one third of chest diameter Stage IIIA limited to spleen or splenic, celiac, or portal nodes and lesions no larger than 6 cm Surgical staging required if: Clinical and imaging findings equivocal Tanner stage IV/V for whom radiotherapy is planned Concurrent registration on protocols POG-8828 (late effects study) and POG- 8829 (epidemiology study) required

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Not specified Hematopoietic: No hematopoietic disease Hepatic: No liver disease Renal: No renal disease Other: No severe organ or system damage or failure No pregnant or nursing women

PRIOR CONCURRENT THERAPY: No prior therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 294 (Actual)
Dates: Start 1996-10; Primary Completion 2004-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
DLCO | 1 year post therapy
  The Wilcoxon test will be used to evaluate whether DLCO values differ between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron K. Tebbi, MD, Study Chair — St. Joseph's Children's Hospital of Tampa; Michael A. Weiner, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (39):
- United States (36):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Tebbi CK, London WB, Friedman D, Villaluna D, De Alarcon PA, Constine LS, Mendenhall NP, Sposto R, Chauvenet A, Schwartz CL. Dexrazoxane-associated risk for acute myeloid leukemia/myelodysplastic syndrome and other secondary malignancies in pediatric Hodgkin's disease. J Clin Oncol. 2007 Feb 10;25(5):493-500. doi: 10.1200/JCO.2005.02.3879. PMID 17290056
- [Background] Schwartz CL, Tebbi CK, Constine LS: Response based therapy for pediatric Hodgkin's disease (HD): Pediatric Oncology Group (POG) protocols 9425/9426. [Abstract] Med Pediatr Oncol 37 (3): A-P219, 263, 2001.
- [Result] Tebbi CK, Mendenhall NP, London WB, Williams JL, Hutchison RE, Fitzgerald TJ, de Alarcon PA, Schwartz C, Chauvenet A. Response-dependent and reduced treatment in lower risk Hodgkin lymphoma in children and adolescents, results of P9426: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2012 Dec 15;59(7):1259-65. doi: 10.1002/pbc.24279. Epub 2012 Aug 21. PMID 22911615
- [Result] Mendenhall NP, Meyer J, Williams J, et al.: The impact of central quality assurance review prior to radiation therapy on protocol compliance: POG 9426, a trial in pediatric Hodgkin's disease. [Abstract] Blood 106 (11): A-753, 2005.